CLINICAL TRIAL: NCT06804018
Title: The Effect of Mandala Colouring Practice on Pregnancy Well-Being, Self-Compassion and Anxiety in Primiparous Pregnant Women: A Randomised Controlled Study
Brief Title: Mandala Colouring: Its Impact on Well-Being, Self-Compassion, and Anxiety in Primiparous Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Abdurrahim UYANIK, Lecturer, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Gaziosmanpasa-AU
Record Dates: First submitted 2025-01-13; First posted 2025-01-31 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Pregnant Women; Women Health; Well Being; Self Compassion; Anxiety
Keywords: Pregnant women; anxiety; well being; self compassion; mandala coloring
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: The data from the study will be examined by an independent statistician. The person doing the analysis will not know the groups. Pregnant women included in the study will later learn which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (pregnant women who will paint mandalas) (Experimental): Each participant in the intervention group will be given 12 different colored felt-tip pens or 12 different colored crayons (whichever the pregnant woman wishes) and mandala pictures taken by the researcher.
  They will be asked to choose the pictures they will color, and the pregnant women will be given mandalas with various patterns.
  They will be asked to color for an average of 20-30 minutes two days a week (on the day and time period they want).
  They will be told that they can do their coloring in an environment they want, that they will not have others do their coloring, and that they will not be called back to the hospital for coloring.
  A reminder message* will be sent by the researcher according to the determined days before each coloring, and photos of the colored mandalas will be sent to the researcher via WhatsApp after coloring.
  Afterwards, it will be explained that the STAI form, the Well-being in Pregnancy Scale, and the Self-Compassion Scale will need to be filled out a to
  Interventions: Other: Mandala coloring
- Control Group (No Intervention): For the control group, the scales and forms will be filled out at the end of the second and fourth weeks. Pregnant women will be asked to fill out the forms at the end of the second and fourth weeks and send them to the researcher via WhatsApp, and they will not be invited to a face-to-face interview again.

INTERVENTIONS:
Other: Mandala coloring — Pregnant women who will paint mandalas
  Arms: Intervention Group (pregnant women who will paint mandalas)

SUMMARY:
Maintaining well-being during pregnancy, reducing anxiety and supporting self-compassion are critical for the health of expectant mothers and the development of the baby. In addition to traditional medicine, alternative therapeutic approaches have been increasingly popular in recent years as a supportive approach during pregnancy. Among these alternative methods, creative activities such as mandala painting have the potential to reduce stress, increase mental focus and provide emotional balance.

H1: There is a difference in well-being, self-compassion and anxiety levels between primiparous pregnant women who painted mandalas and those who did not during pregnancy.

H0: There is no difference in well-being, self-compassion and anxiety levels between primiparous pregnant women who painted mandalas and those who did not during pregnancy.

Sub-Hypotheses of the Study:

H1-1: There is a difference in well-being between primiparous pregnant women who painted mandalas and those who did not during pregnancy.

H1-2: There is a difference in self-compassion levels between primiparous pregnant women who painted mandalas and those who did not during pregnancy.

H1-3: There is a difference in anxiety levels between primiparous pregnant women who painted mandalas and those who did not during pregnancy.

DETAILED DESCRIPTION:
Maintaining well-being, reducing anxiety, and supporting self-compassion during pregnancy are of critical importance for the health of expectant mothers and the development of the baby. In addition to traditional medicine, the use of alternative therapeutic approaches as a support during pregnancy has been increasingly gaining interest in recent years. Among these alternative methods, creative activities such as mandala painting have the potential to reduce stress, increase mental focus, and provide emotional balance (Babouchkina and Robbins, 2015; Stinley et al., 2015; Sandmire et al., 2016; Mo and Ko, 2023; Chen et al., 2024; Şolt Kırca and Dağlı, 2024). However, controlled studies evaluating the effects of mandala painting during pregnancy are limited (Şolt Kırca and Dağlı, 2024). In particular, it seems that the effects of mandala painting on psychological well-being, self-compassion, and anxiety levels in primiparous pregnant women and in the last trimester of pregnancy have not been systematically examined. With these effects, it is thought that mandala painting during pregnancy will be used as a stress management tool recommended by health professionals and will contribute to the field as it can contribute to the emotional well-being of future pregnant women.

Data Collection Tools In collecting the data of the research:

The research data will be collected using the Sociodemographic Characteristics Form, State Anxiety Scale, Pregnancy Well-Being Scale and Self-Compassion Scale Short Form. Sociodemographic Characteristics Form: The form consists of 6 questions in total and includes age, education level, employment status, perceived economic status, number of pregnancies and whether the pregnancy was planned. State Anxiety Scale: The State-Trait Anxiety Inventory (STAI) form developed by Spielberger (1983) is used for adults between the ages of 18-69 and consists of 20 items (state anxiety) measuring the intensity of anxiety as an emotional state (Spielberg, 1983). In order for pregnant women to express their own feelings, they can instantly mark how they feel without spending too much time on any expression, and it is evaluated as 1: not at all, 2: a little, 3: a lot and 4: completely. If no response is given to more than three statements, the completed form is considered invalid and is not scored. Direct statements express negative emotions; reversed statements express positive emotions. When scoring, those with a weight value of 1 are converted to 4, and those with a weight value of 4 are converted to 1. There are ten reverse-coded statements in the state anxiety scale. These are items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. Theoretically, the scores obtained vary between 20 and 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety (Spielberg, 1983). The scale was adapted to Turkish culture by Öner and Le Compte, and a reliability-validity study was conducted. In the Turkish version of the scale, reliability coefficients determined by Cronbach's alpha correlations were found to be between 0.83 and 0.92 (Öner and Le Compte, 1983). Well-Being Scale in Pregnancy: The Turkish validity-reliability study of the scale developed by Alderdice et al. (2015) in 2015 was conducted by Sunay et al. (2022). The Cronbach's alpha reliability coefficient in the original scale is 0.73 (Alderdice et al., 2015). The scale defines the characteristics of well-being measurement during pregnancy and general well-being gives women the opportunity to express their positive and negative feelings and thoughts about their pregnancy. The scale is a six-point Likert-type scale and the responses to the items are scored as "1 = always", "2 = most of the time", "3 = more than half of my time", "4 = less than half of my time", "5 = sometimes", "6 = never". The increase in the average score obtained from the scale indicates that well-being during pregnancy has increased. The scale consists of a total of 12 items and has two subscales: "Positive Affect and Satisfaction" and "Concerns". The Positive Affect and Satisfaction subscale (high scores indicate high positive emotions, positive relationships, and satisfaction with pregnancy and care) consists of 7 items (items 1, 2, 3, 5, 7, 11, and 12). The Concerns subscale (where high scores indicate less anxiety) consists of 5 items (items 4, 6, 8, 9, and 10). The 5 items of the Concerns subscale (items 4, 6, 8, 9, and 10) are calculated by reversing them. The Cronbach's alpha value of the scale was found to be 0.73. The Positive Affect and Satisfaction subscale of the scale was found to be 0.71, and the Concerns subscale was found to be 0.70 (Sunay et al., 2022). Self-Compassion Scale Short Form: The scale developed by Neff (2003) was converted into a short form by Raes, Pommier, Neff, and Van Gucht (2011). The form, whose Turkish validity and reliability study was conducted by Yıldırım and Sarı (2018), consists of a total of 11 questions. It is one-dimensional. The Likert-type scale is marked as 1: never, 2: rarely, 3: sometimes, 4: often, and 5: always. Items 1, 4, 8, 9, 10, and 11 of the scale are reverse-coded. The internal consistency coefficient of the scale was calculated as 0.75. The total scores obtained from the scale indicate that the self-compassion level of the individuals is high (Neff et al., 2003; Yıldırım and Sarı, 2018).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* Being in the last three months of pregnancy (Amelia et al., 2020)
* Getting a State Anxiety Inventory (STAI) score of ≥40
* Having a smartphone and internet connection
* Being willing to participate in the study
* Being spontaneously pregnant
* Not having a diagnosed health risk (diabetes, preeclampsia, fetal anomaly, etc.) in the mother or fetus

Exclusion Criteria:

* Those who do not meet the Inclusion Criteria

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Anxiety Scale | 5 weeks
  The State Anxiety Inventory (STAI-X) will be used to determine the anxiety status of pregnant women.

SECONDARY OUTCOMES:
Well-being | 5 weeks
  The Well-Being in Pregnancy Scale will evaluate pregnant women's cognitive evaluations of their own lives and the frequency and intensity of their positive and negative emotions.

OTHER OUTCOMES:
Self-Compassion | 5 weeks
  Self-compassion levels of primiparous pregnant women will be evaluated with the Self-Compassion Scale Short Form.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Erbaa, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting information: CSR
Supporting Information: CSR